CLINICAL TRIAL: NCT01288456
Title: A Single Centre 30-day Observational Non-randomised Study to Evaluate Preliminary Safety and Efficacy of a Novel Gastric Space Occupying Device as an Aid for Weight Loss
Brief Title: Study to Evaluate Novel Gastric Space Occupying Device
Status: Completed | Type: Observational
Sponsor: Obalon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-1000-0005
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Obesity
Keywords: medical device, space-occupying device
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be an observational, prospective, non-randomized, pilot study to gain initial device experience on a novel space-occupying device in persons who are overweight or obese. No formal hypothesis testing will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21-64 years
2. BMI 27-40 Kg/m2
3. No history of weight reduction of more than 5% of total body weight in the past 6 months

Exclusion Criteria:

1. Have unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity;
2. Be taking chronic aspirin or other non steroidal anti-inflammatory agents, or other medications known to be gastric irritants, and unwillingness to discontinue the use of these concomitant medications, antiarrythmics, anti-anginal medications, anticoagulants or medications for congestive heart failure;
3. Be taking blood pressure medications, unless their blood pressure is controlled and they have been at stable dose for at least 3 months;
4. Have type 1 diabetes or type 2 diabetes requiring oral medications or insulin;
5. History or symptoms of thyroid disease which is not controlled by medication;
6. Have severe renal, hepatic, pulmonary disease or cancer;
7. Past history of gastrointestinal surgery (excluding uncomplicated appendectomy);
8. Have a history of adhesive peritonitis;
9. History or symptoms of esophageal and/or gastric varices;
10. Have history or congenital or acquired GI anomalies (e.g. atresias, stricture, and /or diverticula);
11. History or symptoms of inflammatory bowel disease, such as Chron's disease;
12. History of/ signs and /or symptoms of duodenal or gastric ulcer;
13. Have gastroparesis;
14. Pregnant or breastfeeding or intention of becoming pregnant during the study (if female of childbearing potential);
15. Currently using pharmaceutical agents for weight loss;

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be selected from a community sample that satisfy the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Ortiz, MD, Principal Investigator — Obesity Control Center
Locations (1):
- Obesity Control Center, Tijuana, Estado de Baja California, Mexico